CLINICAL TRIAL: NCT02114073
Title: Comparison of Effect of Cyclosporine Ophthalmic Emulsion 2% and Betamethasone Eye Drop on Intraocular Pressure, Conjunctival Hyperemia and Subjective Dry Eye Symptoms Following Trabeculectomy in Open Angle Glaucoma Patients
Brief Title: Comparison of Effect of Postoperative Cyclosporine A 2% Ophthalmic Emulsion and Betamethasone Eye Drop on Surgical Success of Trabeculectomy Procedure
Acronym: BCATS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ramin Daneshvar, MD, Dr. Ramin Daneshvar, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUMS-911251; IRCT138706111154N1 (Other: Iranian Registery of Clinical Trial)
Record Dates: First submitted 2014-04-06; First posted 2014-04-15 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Glaucoma, Open Angle
Keywords: glaucoma; trabeculectomy; cyclosporine; betamethasone
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Cyclosporine; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine (Experimental): In the first postoperative day following a standard, fornix-based trabeculectomy, ophthalmic emulsion of Cyclosporine A, 2%, every 4 hours for the first postoperative week and every 6 hours for the next 3 weeks will be prescribed for the patients.
  Interventions: Drug: Cyclosporine
- Betamethasone (Active Comparator): In the first postoperative day following a standard, fornix-based trabeculectomy, betamethasone eye drop, every 4 hours for the first postoperative week and every 6 hours for the next 3 weeks will be prescribed for the patients.
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Cyclosporine — In study arm, ophthalmic emulsion of cyclosporine A 2% will be prescribed in postoperative phase.
  Other Names: Cyclosporine A (Sina Darou)
  Arms: Cyclosporine
Drug: Betamethasone — In control arm, betamethasone eye drop will be prescribed in postoperative period.
  Other Names: Betasonate (Sina Darou)
  Arms: Betamethasone

SUMMARY:
Glaucoma is one of the leading causes of blindness worldwide and trabeculectomy is the most commonly performed operation to slow-down the disease progression. In this study, we compare the effect of topical cyclosporine A and betamethasone eye drops on the postoperative course and surgical success of trabeculectomy.

DETAILED DESCRIPTION:
Trabeculectomy is still the most popular filtering surgery for glaucomatous patients. In this type of surgery, postoperative care and management is highly important for surgical success. A principle component of postoperative regimen is anti-inflammatory medications. However, corticosteroid eye drops, the most frequently used agents, have some side effects, including raising intraocular pressure.

Cyclosporine A could be an interesting alternative, because not only it has acceptable anti-inflammatory effect and could reduce some ocular surface problems, but also it has minimal direct effect on intraocular pressure. In this study, we will compare the effect of topical cyclosporine A and betamethasone on surgical outcome and postoperative course of trabeculectomy patients.

The study is a prospective study to compare the effect of topical betamethasone and cyclosporine A on postoperative findings of glaucoma patients, undergoing trabeculectomy surgery.

In this study, trabeculectomy patients, who fulfill the study criteria, will be randomized to either study group and follow-up visits will be done in a masked fashion. In each visit, a detailed history taking and eye examination will be done by an examiner unaware of study group. A third party would do data control for patient safety. At the conclusion of the study, the data of the two groups would be compared. All human research ethical codes are strictly respected and the Ethical Committee of the University has an ongoing inspection on all study steps.

We hypothesize that cyclosporine A could provide better inflammation and intraocular pressure control and may enhance surgical success rate. However, our null hypothesis is that the result in study groups will not differ statistically significantly.

ELIGIBILITY:
Inclusion Criteria:

* POAG patient with insufficient IOP control on maximal tolerable medical therapy (MTMT), undergoing primary trabeculectomy with MMC augmentation.

Exclusion Criteria:

* Age <20 years
* History of previous ocular surgery in the same eye;
* Candidate for combined surgery;
* Pregnancy;
* Breast feeding;
* Monocular subject;
* Allergy to any topical antiglaucoma medication or cyclosporine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure (IOP) | Up to 6 months after surgery
  Each month following trabeculectomy, intraocular pressure will be measured using Goldmann Applanation Tonometer.
Bleb morphology | Up to 6 months after surgery
  Bleb morphology according to IBAGS grading system, based on clinical examination and slit-lamp photography.
Subjective dry eye symptoms | Up to 6 months after surgery
  Subjective symptoms of dry eye, reported by patients, and gathered using a standardized questionnaire.

SECONDARY OUTCOMES:
Surgical success rate | 6 month after surgery
  The surgical success rate of trabeculectomy in each study arm.
Complications | Up to 6 months after surgery
  Any complication observed during study period, reported by patient or examiner.
Visual acuity | Up to 6 months after surgery
  LogMAR visual acuity, measured on every postoperative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Daneshvar, MD, MSc, Principal Investigator — Eye Research Center, Cornea Research Center, Mashhad University of Medical Sciences
Locations (1):
- Khatam Eye Hospital, Mashhad, Khorasan Razavi, Iran